CLINICAL TRIAL: NCT02440581
Title: Renal Osteodystrophy: A Fresh Approach
Brief Title: Renal Osteodystrophy: An Individual Management Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartmut Malluche, MD (Other)
Collaborators: Wright State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Hartmut Malluche, MD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0976-F6A; R01DK080770 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Alendronate; Teriparatide; Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control, low turnover (No Intervention): No intervention in low turnover osteoporosis control group.
- Treatment, low turnover (Experimental): Low turnover osteoporosis group treated with teriparatide and cinacalcet.
  Interventions: Drug: Teriparatide; Drug: Cinacalcet
- Control, high turnover (No Intervention): No intervention in high turnover osteoporosis control group.
- Treatment, high turnover (Experimental): High turnover osteoporosis group treated with alendronate.
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate
  Arms: Treatment, high turnover
Drug: Teriparatide
  Arms: Treatment, low turnover
Drug: Cinacalcet
  Arms: Treatment, low turnover

SUMMARY:
Renal osteodystrophy (ROD) represents the bone histologic abnormalities resulting from loss of renal function. It starts early during the loss of kidney function and is seen in virtually all chronic end stage kidney disease patients on dialysis (CKD-5D). A major component of ROD is bone loss leading to chronic kidney disease (CKD) associated osteoporosis. Debilitating hip fractures occur in patients with CKD at a rate 4.4 times higher than in the general population, with associated high costs, morbidity and an annual mortality of 64%. CKD osteoporosis is distinctly different from post-menopausal osteoporosis. Presently, no uniformly accepted CKD osteoporosis treatment protocol exists because of challenges related to racially specific bone turnover states. Therefore, most physicians are reluctant to treat this disorder despite the profound impact on health and quality of life, and its association with vascular calcifications. These vascular calcifications confer an increased risk for cardiovascular events which are the major cause of the over 20% annual mortality rate in CKD-5D patients.

The goal of the proposed controlled randomized study is to test the concept that CKD osteoporosis can be successfully treated when treatment is individualized by patients' turnover status. The study will demonstrate that reversal of bone loss can be achieved by increasing bone formation in low turnover patients, and by reducing bone resorption in normal or high turnover patients. A second aim of this study is to provide new information whether these treatments will also retard progression of vascular calcifications. Blood tests measuring FGF23, indicators of Wnt pathway activity, bone resorption and formation will be followed to understand potential mechanisms and to evaluate their usefulness for prediction of changes in bone mass and vascular calcifications.

CKD-5D patients with established osteoporosis will be enrolled into one of two treatment arms based on bone turnover status. Each arm will be adaptively randomized by race, age and gender into treatment or control groups. In the low turnover arm, teriparatide combined with cinacalcet will be given, and in the normal or high turnover arm, alendronate will be administered. Bone mineral density will be measured at baseline and after one year of treatment by quantitative computed tomography. Calcifications of the coronaries, aorta and heart valves will also be measured at the same times by multi-detector computed tomography.

If this proof-of-concept study is successful, it will offer a heretofore unavailable treatment for osteoporosis in CKD-5D patients thus changing the prevailing clinical practice paradigm. This will provide immediate benefit to CKD patients by reducing fracture risk, bone pain, and cardiovascular risk, while greatly improving their quality of life. These improvements will also convey major socioeconomic benefits by decreasing the high associated treatment costs. The proposed study is highly relevant to the National Institute of Diabetes and Digestive and Kidney Diseases' mission of disseminating science-based information to improve the health and quality of life for patients with endocrine, metabolic and kidney diseases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years or older;
* Chronic maintenance dialysis of at least 3 months' duration;
* Osteoporotic by DXA of either spine or total hip (Women: post-menopausal or age ≥ 50 with T-score ≤ -2.5; Men: age ≥ 50 with T-score ≤ -2.5; All others, Z-score ≤ -2.5);
* Mental competence;
* Willingness to participate in the study;
* Normal serum calcium.

Exclusion Criteria:

* Pregnancy or breast feeding;
* Incarceration;
* Systemic illnesses or organ diseases that may affect bone (except type 1 or type 2 diabetes mellitus);
* Clinical condition that may limit study participation (e.g., unstable angina, respiratory distress, infections).
* Chronic alcoholism and/or drug addiction;
* Known Paget 's disease of bone;
* Prior external beam or implant radiation therapy involving the skeleton;
* More than 3 computed tomography (CT) scans in the prior 12 months (to avoid excessive radiation exposure);
* Participation in a study of an investigational drug during the past 90 days;
* Planning to move out of the area within 1 year of the study;
* On active transplant list;
* BMD t-score of the radius less than -3.5 by DXA (to avoid the known potential negative effects of teriparatide treatment on BMD of the radius);
* Planned or anticipated oral surgery within the next 12 months;
* Inability to stand or sit upright for at least 30 minutes;
* Abnormalities of the esophagus which delay esophageal emptying such as stricture or achalasia;
* Treatment within last 6 months with drugs that may affect bone metabolism including bisphosphonates and teriparatide (except for treatment with calcitriol, vitamin D analogs and/or calcimimetics);
* Current treatment with medicines containing digoxin or warfarin;
* Calcidiol level below the normal range. (The current routine clinical practice in our dialysis clinics is to check calcidiol status twice yearly and supplement with vitamin D according to serum calcidiol levels. It is therefore unlikely that a substantial number of patients will be excluded due to this exclusion criterion.)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Malluche, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment, Low Turnover: Low turnover osteoporosis group treated with teriparatide and cinacalcet.
  Teriparatide
  Cinacalcet
- Treatment, High Turnover: High turnover osteoporosis group treated with alendronate.
  Alendronate
Period: Overall Study
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover
Started | 37 | 24 | 50 | 30
Completed | 32 | 13 | 37 | 16
Not Completed | 5 | 11 | 13 | 14
Not completed — Death | 0 | 0 | 7 | 5
Not completed — Transplanted | 1 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 4 | 11 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover | Total
Number analyzed (Participants) | 37 | 24 | 50 | 30 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 12 | 32 | 17 | 89
  >=65 years | 9 | 12 | 18 | 13 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.68 (1.95) | 62.67 (2.83) | 59.14 (1.73) | 59.83 (2.28) | 61.035 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 23 | 12 | 60
  Male | 21 | 15 | 27 | 18 | 81
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 10 | 9 | 24 | 6 | 49
  White | 27 | 15 | 26 | 24 | 92
Region of Enrollment [Number; unit: participants]
  United States | 37 | 24 | 50 | 30 | 141

OUTCOME MEASURES:

1. Primary Outcome: Change in Quantitative Computed Tomography (QCT) Bone Mineral Density of the Hip
Description: At one year the investigators will asses bone mass using QCT of the total hip and compare one year changes in bone mass between the treatment and control groups.
Time Frame: One Year (at baseline and one year)
Measure: Mean (Standard Error); unit: g/cm^3
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover
Number analyzed (Participants) | 37 | 24 | 50 | 30
g/cm^3 | -10.71 (4.73) | 5.72 (4.74) | -3.52 (3.36) | .2 (5.67)
Statistical Analysis 1: Comparison: Control, Low Turnover vs Treatment, Low Turnover vs Control, High Turnover vs Treatment, High Turnover; Test type: Other — T-tests; p = .443, t-test, 2 sided

2. Secondary Outcome: Change in Coronary Artery Calcifications by Multiple Detector Computed Tomography (MDCT)
Description: At one year the investigators will asses differences between the treatment and control groups in changes in Coronary Artery Calcifications by MDCT. 1 Yr. Change in Sqrt CAC Vol.
Time Frame: One year (at baseline and one year)
Measure: Mean (Standard Error); unit: Hounsfield Unit
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover
Number analyzed (Participants) | 37 | 24 | 50 | 30
Hounsfield Unit | 2.78 (1.51) | 4.48 (1.83) | 4.97 (1.89) | 3.47 (1.28)
Statistical Analysis 1: Comparison: Control, Low Turnover vs Treatment, Low Turnover vs Control, High Turnover vs Treatment, High Turnover; Test type: Other — T-tests; p = .490, t-test, 2 sided

3. Secondary Outcome: Change in Serum Biochemical Bone Markers of Bone Activity - Parathyroid Hormone (PTH)
Description: Bone markers of bone activity tracked over time for changes.1 Yr. Change in PTH
Time Frame: 1 Year (at baseline and one year)
Population: 1 Yr. Change in PTH
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover
Number analyzed (Participants) | 37 | 24 | 50 | 30
pg/ml | 89 (32.3) | 379 (118.6) | -125 (81.2) | -240 (126.5)
Statistical Analysis 1: Comparison: Control, Low Turnover vs Treatment, Low Turnover vs Control, High Turnover vs Treatment, High Turnover; Test type: Other — T-tests; p < .001, t-test, 2 sided

4. Secondary Outcome: Change in Serum Biochemical Bone Markers of Bone Activity - Bone-specific Alkaline Phosphatase (BSAP)
Description: Bone markers of bone activity tracked over time for changes.1 Yr. Change in BSAP
Time Frame: 1 year (at baseline and one year)
Population: 1 Yr. Change in BSAP
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover
Number analyzed (Participants) | 37 | 24 | 50 | 30
pg/ml | .61 (3.683) | -1.01 (4.616) | -8.92 (6.121) | -10.36 (5.522)
Statistical Analysis 1: Comparison: Control, Low Turnover vs Treatment, Low Turnover vs Control, High Turnover vs Treatment, High Turnover; Test type: Other — T-Tests; p = .083, t-test, 2 sided

5. Secondary Outcome: Change in Serum Biochemical Bone Markers of Bone Activity - Fibroblast Growth Factor 23 (FGF23)
Description: Bone markers of bone activity tracked over time for changes. 1 Yr. Change in FGF-23
Time Frame: 1 Year (at baseline and 1 year)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover
Number analyzed (Participants) | 37 | 24 | 50 | 30
pg/ml | 985 (1611) | 326 (1114) | 3337 (1427) | 607 (467)
Statistical Analysis 1: Comparison: Control, Low Turnover vs Treatment, Low Turnover vs Control, High Turnover vs Treatment, High Turnover; Test type: Other — T-tests; p = .283, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Years 1-5
Arm/Group | Control, Low Turnover | Treatment, Low Turnover | Control, High Turnover | Treatment, High Turnover
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/24 | 7/50 | 5/30
Serious Adverse Events (participants affected / at risk) | 16/37 | 10/24 | 21/50 | 16/30
Other Adverse Events (participants affected / at risk) | 16/37 | 16/24 | 19/50 | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control, Low Turnover (N=37) | Treatment, Low Turnover (N=24) | Control, High Turnover (N=50) | Treatment, High Turnover (N=30)
Acute blood loss anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Eliquis-associated bleeding (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Scrotal hematoma (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
A. fib (Cardiac disorders) | 1 | 0 | 0 | 0
Heart attack (Cardiac disorders) | 0 | 0 | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0 | 0
Orbital cellulitis (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Blood in stool (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulitis, hypoglycemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GI bleed (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea/vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 5 | 7 | 0 | 0
Fatigues/weakness (General disorders) | 0 | 0 | 0 | 1
Generalized weakness/fall (General disorders) | 1 | 0 | 0 | 0
Weakness (General disorders) | 0 | 4 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1
Flu (Infections and infestations) | 0 | 0 | 1 | 0
Flu A (Infections and infestations) | 1 | 0 | 0 | 0
Flu/bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Foot Infection (Infections and infestations) | 0 | 0 | 0 | 1
Left foot infection (Infections and infestations) | 0 | 0 | 0 | 1
Mono/RSV (Infections and infestations) | 0 | 0 | 1 | 0
MRSA bacteremia (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 1
Sepsis s/p UTI (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Femur fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Left foot fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Left hand fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Left hip fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Left hip replacement s/p fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Left knee pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar/cervical stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pinched Nerve (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Right hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Right leg fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Possible thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Altered mental status (Nervous system disorders) | 0 | 0 | 0 | 1
Altered mental status and weakness (Nervous system disorders) | 0 | 1 | 0 | 0
Decreased LOC (Nervous system disorders) | 0 | 1 | 0 | 0
Slurred speech (Nervous system disorders) | 0 | 1 | 0 | 0
Blocked PD catheter (Renal and urinary disorders) | 0 | 0 | 1 | 0
Fluid overload (Renal and urinary disorders) | 1 | 1 | 2 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Polycystic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
UTI (Renal and urinary disorders) | 0 | 2 | 0 | 1
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Pneumonia with SOA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia/bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory/cardiac arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
SOA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2
SOA, chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
SOA/fluid overload, hyperglycemia, pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
URI with ascites (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Right foot ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Right nephrectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Scheduled sinus surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0
AV graft infection (Vascular disorders) | 1 | 0 | 0 | 0
CVA (Vascular disorders) | 0 | 1 | 0 | 0
Fistula repair (Vascular disorders) | 0 | 0 | 0 | 1
Left great toe amputation (Vascular disorders) | 0 | 2 | 0 | 0
Left metatarsal amputations (Vascular disorders) | 1 | 0 | 0 | 0
Left third toe gangrene (Vascular disorders) | 0 | 1 | 0 | 0
Occluded fistula (Vascular disorders) | 0 | 2 | 0 | 0
Right transmetatarsal amputation (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control, Low Turnover (N=37) | Treatment, Low Turnover (N=24) | Control, High Turnover (N=50) | Treatment, High Turnover (N=30)
Left leg contusion (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Possible blood clot in leg (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Chest pain (Cardiac disorders) | 0 | 1 | 1 | 1
Elevated BP during dialysis (Cardiac disorders) | 0 | 0 | 1 | 0
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
SVT (Cardiac disorders) | 0 | 0 | 0 | 1
Ruptured right tympanic membrane (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Increased PTH (Endocrine disorders) | 0 | 0 | 0 | 1
Left red eye (Eye disorders) | 0 | 1 | 0 | 0
Red, painful right gr toe (Eye disorders) | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal cramps, nausea/vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain, nausea/vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 2
N/V, diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea/coughing (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea/diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea/vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea/vomiting, lightheadedness (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea/vomiting/ (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Reflux/vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach virus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1
Fatigue, muscle ache (General disorders) | 0 | 0 | 1 | 0
Front tooth removal (General disorders) | 0 | 1 | 0 | 0
Headache (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Poor appetite (General disorders) | 1 | 0 | 0 | 0
Right side pain (General disorders) | 2 | 0 | 0 | 0
Weakness (General disorders) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Fever (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Left arm infection (Infections and infestations) | 0 | 0 | 0 | 1
Left lower extremity wound (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinus infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 1 | 1
Frequent falls (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Right toenail avulsion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dizziness (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Weight loss (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bilateral heel pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bilateral leg aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bilateral leg pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Bilateral leg weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bilateral shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Bilateral thigh pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
BL wrist pain and right thumb pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bruised ribs (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Carpal tunnel (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Immobility (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Left arm pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Left foot pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Left foot/ankle pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Left forearm pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Left hip injury (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Left hip pain/weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Left knee pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Left rib fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Left rib/abdominal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Left side pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Leg aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Leg weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Low back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Low back/hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Right ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Right arm swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Right carpal tunnel (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Right foot pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Right hip pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Right knee pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Right rib pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Right wrist synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Second ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Swelling at lower extremity prosthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Appetite suppression (Nervous system disorders) | 0 | 1 | 0 | 0
BL neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Forgetfulness (Nervous system disorders) | 0 | 1 | 0 | 0
Forteo pen ran out early (Product Issues) | 0 | 0 | 1 | 0
Teriparatide injection issues (Product Issues) | 0 | 0 | 1 | 0
Possible UTI (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
UTI (Renal and urinary disorders) | 0 | 2 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Breathing difficulty (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough/congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
SOA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
URI (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Abscess on bottom (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Bottom wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Foot ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Plantar wart right gr toe (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Right foot wound (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Scalp sores (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Bed bugs (Social circumstances) | 0 | 0 | 0 | 1
PD catheter revision (Surgical and medical procedures) | 0 | 0 | 1 | 0
Vascular Disorders (Surgical and medical procedures) | 0 | 0 | 0 | 0
Poor circulation in left foot (Surgical and medical procedures) | 0 | 1 | 0 | 0
Splenic artery aneurysm (Surgical and medical procedures) | 0 | 1 | 0 | 0
Thrombosed AV fistula (Surgical and medical procedures) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT02440581/Prot_SAP_ICF_000.pdf